CLINICAL TRIAL: NCT01554267
Title: The Use of Laser-Assisted Indocyanine Green Dye Angiography to Predict Intraoperative Mastectomy Skin Flap Viability During Breast Reconstruction
Brief Title: The Use of Laser-Assisted Indocyanine Green Dye Angiography to Predict Mastectomy Skin Flap Viability
Acronym: ICG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Stony Brook University (Other)
Responsible Party: Principal Investigator, Duc T Bui, MD, Associate Professor of Surgery, Stony Brook University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 127891
Record Dates: First submitted 2012-03-12; First posted 2012-03-14 (Estimated); Last update posted 2014-05-13 (Estimated); Status verified 2014-05

CONDITIONS: Breast Cancer; Breast Reconstruction; Mastectomy
Keywords: Mastectomy skin flap necrosis; Breast reconstruction; Indocyanine Green Dye
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mastectomy Skin Flap SPY Excision (Experimental): Single arm study where areas of necrosis predicted by Laser-Assisted Indocyanine Green Dye Angiography (SPY system) will be excised intraoperatively during breast reconstruction surgery.
  Interventions: Device: Laser-Assisted ICG Dye Angiography (SPY System)

INTERVENTIONS:
Device: Laser-Assisted ICG Dye Angiography (SPY System) — 7.5-10mg of ICG dye will be injected at 2 different time points during breast reconstruction with the assistance of the SPY system to determine areas of skin with poor blood flow. These areas are excised during the operation in order to decrease postoperative complications including mastectomy skin flap necrosis and reconstruction failure.
  Other Names: Lifecell SPY System; Novadaq SPY System

SUMMARY:
In the investigators previous study of 51 breast reconstructions (32 patients), we compared three different assessments of vascular perfusion of tissue; clinical judgment, fluorescein dye angiography (FDA) and laser-assisted indocyanine green dye angiography (ICG). Because tissue with poor perfusion becomes necrotic and can compromise the success of breast reconstruction, it is important that tissue with poor perfusion be removed at the time of the reconstructive surgery. However, it is also important to remove the least amount of potentially necrotic tissue as possible so that the breast reconstruction is not compromised by lack of skin. Therefore finding the best way to assess potentially necrotic tissue is a vital clinical question. In the initial study the 3 different assessment methods which were made at the time of surgery were compared to the subsequent development of necrotic tissue.

In the initial study, clinical judgment was the basis for determining the tissue removed because it had the potential to become necrotic. The investigators collected data with the FDA system and ICG system, but this data was not used in making the clinical decisions. The study followed the progression of tissue to overt necrosis and this clinical outcome was then compared to the predictions made by the three different assessment strategies. The investigators found that clinical judgment failed to detect tissue which subsequently became necrotic in 21 out of 51 instances for a failure rate of 41%. The FDA system predicted larger areas of potentially necrotic tissue than clinical judgment, but was found to over-predict the area that became necrotic by 82% - 88% (88% if all cases were included and 82% if only those cases which subsequently developed necrosis were included). Although the ICG system is similar to the FDA system in that a dye is used to assess perfusion, the ICG system has enhanced software which improves the estimated perfusion. The ICG system provided 90% sensitivity and 100% specificity in the predicted vs. actual necrotic tissue at specific absolute perfusion units values.

Hypothesis: Using the values of absolute perfusion units discovered in the previous study and implementing its use in the operating room will decrease all-inclusive necrosis rates to below 10%, reflecting a 31% decrease in the investigators necrosis rate.

DETAILED DESCRIPTION:
The investigators current rate of the development of all-inclusive mastectomy skin necrosis was approximately 41%. This means that current methods of clinical assessment fail to identify regions of mastectomy skin with poor blood flow that lead to necrosis in 41% of patients. The investigators know that using the SPY imaging system is more sensitive for necrosis than clinical assessment. With SPY Q analysis the investigators hope to obtain 90% sensitivity, 100% specificity at absolute perfusion unit values identified in the previous study. The investigators do not anticipate obtaining a 0% all-inclusive necrosis rate but do believe they can eliminate all clinically significant necrosis that would result in operative debridement or removal of implant. The less severe forms of necrosis including epidermolysis and incisional necrosis are self-limiting and usually do not require invasive interventions.

ELIGIBILITY:
Inclusion Criteria:

1. Being scheduled for unilateral or bilateral mastectomy (prophylactic or for the treatment of cancer) followed by breast construction using a Tissue Expander
2. Consent to participation in the study.

Exclusion Criteria:

1. Refusal to consent to participation in the study
2. Inability to tolerate the administration of indocyanine green dye due to iodine allergy
3. A positive pregnancy test during preoperative evaluation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-01 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
Mastectomy Skin Flap Necrosis | 30 days postop
  All-inclusive mastectomy skin flap necrosis including: epidermolysis, partial/superficial necrosis, and full-thickness necrosis.

SECONDARY OUTCOMES:
Infection | 30 days postop
  Superficial, Deep or Organ space surgical site infection as defined by the CDC. Patients treated with oral or IV antibiotics will be documented, including patients who have loss of implant due to infection.
Wound Dehiscence or Implant Extrusion | 30 days postop
  Wound breakdown and exposure of acellular dermal matrix and implant will be documented.
Seroma/Hematoma | 30 days postop
  Any evidence of seroma/hematoma will be documented and be documented based on requirement of a surgical intervention or observation.
Removal or Loss of Implant | 30 days postop
  Patients who require removal of their implants will be documented along with the primary cause of their loss of implant.

CONTACTS AND LOCATIONS:
Overall Officials: Duc T Bui, MD, Principal Investigator — Stony Brook University; Brett T Phillips, MD, Study Director — Stony Brook University
Locations (1):
- Stony Brook University, Stony Brook, New York, United States